CLINICAL TRIAL: NCT00793988
Title: Vibration-Assisted Anaesthesia: A Randomised Controlled Trial to Investigate Whether Vibration Reduces the Pain of Anaesthetic Injection in Eyelid Surgery
Brief Title: Vibration-Assisted Anaesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Peter Dolman MD, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H08-02244
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Dermatochalasis; Blepharoptosis
Keywords: vibration; local anaesthesia; ptosis surgery; blepharoplasty; Upper eyelid surgery; dermatochalasis +/- blepharoptosis
MeSH Terms: conditions — Cutis Laxa; Blepharoptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Group receiving vibration-assisted anaesthesia
  Interventions: Procedure: Vibration-assisted anaesthesia
- 2 (Placebo Comparator): Group receiving switched-off vibrating device
  Interventions: Procedure: Switched-off vibrating device

INTERVENTIONS:
Procedure: Vibration-assisted anaesthesia — All anaesthetic injections will consist of xylocaine 1% with 1:100,000 adrenaline and will be administered through a short 30 Gauge needle at a constant slow speed at multiple (6-7) sites along the upper lid by a single oculoplastic consultant.
  The vibration device and placebo will be operated by a single oculoplastics fellow. The vibrating device / placebo will be placed on the middle of the forehead 1 cm above the mid-brow point 1 second before the anaesthetic injection is commenced. It will be lifted off the skin every time the injection needle exits the skin and it will be replaced on the same point 1 second before the needle reenters the skin at a new injection site.
  Arms: 1
Procedure: Switched-off vibrating device — The placebo consists of a switched-off vibrating device applied to the test site and a second identical switched-on vibrating device held close (but not touching) the first, which will therefore make the same sound. Care will be taken to ensure that the devices are out of the participants' view. The test and placebo will be randomly assigned to either the first or second eyelid; the right eyelid will be injected first in all patients, as is our routine practice.
  Arms: 2

SUMMARY:
Aim of study is to investigate whether a small, non-invasive vibrating device applied to the forehead during local anaesthetic administration reduces the pain of the injection.

DETAILED DESCRIPTION:
Purpose:

To carry out a prospective randomised controlled clinical trial to compare the efficacy of vibration in reducing the pain of local anaesthetic injections into the upper eyelid.

Hypothesis:

Vibration of the adjacent soft tissue reduces the pain of anaesthetic injections in upper eyelid surgery.

Justification:

In many surgical procedures performed under local anaesthetic, the most frightening and painful aspect of the procedure for patients is the anaesthetic injection, and various techniques have been advocated to address this.

Explaining to the patient beforehand what to expect, talking during the injection and hand-holding can be helpful in relaxing and distracting some patients; however, this alone is unlikely to be sufficient to relieve the pain of the injection in most cases.

Simple measures that reduce the pain of anaesthetic injection and are widely practised include administering the injection slowly and using a fine-bore needle (30 Gauge). Other techniques that have been shown to be effective include warming or buffering the local anaesthetic [1-6]. The use of 0.9% bacteriostatic saline solution in conjunction with lidocaine has been demonstrated to significantly reduce patients' perceived pain during the injection and operative procedure in eyelid surgery [7].

Cooling the skin immediately prior to treatment has been shown to reduce the pain of dermatological laser procedures [8-10] although this might be difficult to perform around the eyes because of the risk of injuring the cornea. Similarly, topical anaesthetic agents, such as EMLA (eutectic mixture of local anaesthetics) cream, which are applied to the skin one hour prior to injection are commonly employed for use on the limbs of infants and children but are not safe for use around the eyes since inadvertent ocular application causes corneal de-epithelisation [11].

Sedative agents, such as midazolam may be useful in anxious patients, but this requires the input of an anaesthetist and it is often difficult to finely control the level of sedation; it is usually preferable not to have patients sedated during eyelid surgery when patient cooperation is required intra-operatively to assess the height of the eyelids, for example in ptosis surgery.

Vibration, pinching or the application of pressure has long been recognised as a method of reducing concurrent pain. In 1965 Melzack and Wall published their gate control theory of pain in which they asserted that the stimulation of vibration or touch receptors in the skin causes stimulation of inhibitory interneurons in the spinal cord which can in turn inhibit the transmission of pain signals to the brain.[12] Other hypotheses to explain the mechanism of action of hyper-stimulatory anaesthesia relate to an acupuncture-type effect, distraction, self-hypnosis or suggestion in credulous patients, but the consensus view is that the gate theory is at least in part relevant in the explanation. [13, 14] There is much anecdotal evidence of the use of such techniques to reduce the pain of anaesthetic injection, mostly in dentistry and dermatology [14-17] but there is a dearth of evidence from randomised controlled trials; a recent randomised clinical study in paediatric dental patients found that counterstimulation, using the thumb to vibrate the soft tissue adjacent to the injection site, in conjunction with a distraction exercise (lifting alternate legs in turn) effectively reduced the pain of anaesthetic injection. [18] There are no reports of vibration anaesthesia in an ophthalmic setting.

Objectives:

The aim of this study is to carry out a randomised controlled study to investigate the effect of vibration-assisted anaesthesia in reducing the pain of local anaesthetic injection for upper eyelid surgery.

A pilot study carried out prior to this proposal investigated the feasibility and potential benefits of this trial with very promising results.

Prior to the pilot study various different vibrating devices (including tuning forks of two different frequencies, an electric toothbrush (with a soft rubber cap instead of a brush head) and several models of handheld massagers) were trialled by the investigators on themselves and colleagues to find the optimal device. Once the preferred instrument (a handheld massager) was selected it was tested on various different sites (including midbrow, mid forehead, over the supraorbital notch, lower eyelid, thumbnail and palm) by verbally-consenting patients undergoing bilateral eyelid surgery in order to find the optimal site. The patients received the massager during injection on one side but not the other (some first eye, some second eye) and were asked to verbally rate the pain scores of the two sides. The consensus opinion was that the greatest effect was produced by vibration in the middle of the forehead.

The pilot study was then conducted on 15 verbally consenting patients undergoing bilateral upper eyelid surgery; during the anaesthetic injection on one side they received vibration and the other side received no vibration. Patients were asked to rate the pain of both injections verbally on a scale of 0 to 10. 12 out of 15 patients found the anaesthetic injection on the side with vibration to be less painful than the side without.

Research Methods:

The study will be a prospective, interventional, randomised, controlled clinical trial.

All patients who fit the inclusion criteria will be offered participation in the trial on the day their surgery is booked. They will be given an information leaflet about the trial, explaining the aim of the study without describing the effect of the vibrating device and placebo in order to reduce the risk of biasing their perception. They will be advised that non-participation will not affect their care in anyway.

The intervention is of no risk to the patient and will not affect the surgical procedure in any way. Any questions that the patient has will be addressed beforehand and they will be required to sign a consent form prior to inclusion in the trial.

They will be advised beforehand that they will be required to verbally rate their pain score on a scale of 0 to 10 immediately after both sides have been anaesthetised, with 0 being no pain and 10 being the worst imaginable pain.

All participants included in the study will undergo bilateral surgery and will therefore act as their own controls: the vibrating device will only be applied whilst the anaesthetic is being injected into one side; a placebo will be applied to the other side. The placebo consists of a switched-off vibrating device applied to the test site and a second identical switched-on vibrating device held close (but not touching) the first, which will therefore make the same sound. Care will be taken to ensure that the devices are out of the participants' view. The test and placebo will be randomly assigned to either the first or second eyelid; the right eyelid will be injected first in all patients, as is our routine practice. Computer-generated sequential binary randomisation will be used. Allocation will be concealed from the surgeon until immediately prior to the anaesthetic injection.

All anaesthetic injections will consist of xylocaine 1% with 1:100,000 adrenaline and will be administered through a short 30 Gauge needle at a constant slow speed at multiple (6-7) sites along the upper lid by a single oculoplastic consultant.

The vibration device and placebo will be operated by a single oculoplastics fellow. The vibrating device / placebo will be placed on the middle of the forehead 1 cm above the mid-brow point 1 second before the anaesthetic injection is commenced. It will be lifted off the skin every time the injection needle exits the skin and it will be replaced on the same point 1 second before the needle reenters the skin at a new injection site.

Patients' verbal pain scores will be elicited and documented immediately by the oculoplastic fellow.

Statistical analysis:

From a pilot study which involved asking 15 patients undergoing upper eyelid surgery to rate the pain they experienced on injection of the local anaesthetic on a scale of 0 to 10, we found pain scores to be sufficiently Normal for an estimation of the sample size to be based on a Normal distribution.

A comparison of the pain scores between the side receiving vibration and the side receiving placebo will be made using the paired t-test.

Planned sample size On a scale of 0 to 10 a difference in pain score of 1.5 may be considered to be clinically significant. The power calculation for a paired t-test with 90% power and p=0.05 demonstrated that a sample size of 80 patients to be more than sufficient to detect a significant difference.

The results will be submitted for publication in a peer-reviewed ophthalmological journal and presentation at international ophthalmological meetings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 16 years) undergoing bilateral upper eyelid surgery under local anaesthetic who have given fully informed consent to be in the trial

Exclusion Criteria:

* Age less than 16 years
* Previous upper eyelid surgery

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Patients' verbal pain scores will be elicited and documented immediately by the oculoplastic fellow. | Immediately

CONTACTS AND LOCATIONS:
Overall Officials: Peter Dolman, MD, Principal Investigator — University of British Columbia
Locations (1):
- Eye Care Centre (operating rooms), Vancouver, British Columbia, Canada